CLINICAL TRIAL: NCT06921707
Title: SC2i-WounDx-001-WounDx™ Pilot Trial: Proof of Concept Feasibility for the Clinical Operations of WounDx™ in Aiding Clinicians Identify Wounds That Are Ready For Surgical Closure
Brief Title: Pilot Trial for WounDx™ Clinical Decision Support Tool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Duke University (Other); University of Alabama at Birmingham (Other); Brooke Army Medical Center (U.S. Federal Agency); Grady Memorial Hospital (Other); Indiana University Health (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00117915; HU0001-23-2-0030 (Other: Department of Defense)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Wounds; Wounds and Injuries; Extremity Injury; Traumatic Wounds and Injuries; Amputation, Traumatic/Surgery; Amputation, Wound; Open Fracture Wounds
Keywords: Wounds; Extremity Injury; Clinical Decision Support Tool; Delayed Wound Closure; Cytokine Biomarkers; Wound Effluent; Traumatic Extremity Wounds
MeSH Terms: conditions — Wounds and Injuries | interventions — Standard of Care; Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: The trial design, is a parallel group randomized controlled study where participants are randomized to either the control group that receives the standard of care of serial wound irrigation, Negative Pressure Wound Therapy, and surgical debridement with the attending clinician determining if a wound is ready to close, or the interventional group that receives standard of care plus the WounDx™ report to augment the clinicians' judgment regarding the wounds readiness to close.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard of Care (Active Comparator): This is the control group that receives the standard of care of serial wound irrigation, Negative Pressure Wound Therapy, and surgical debridement with the attending clinician determining if a wound is ready to close.
  Interventions: Procedure: Standard of Care (SOC)
- WounDx (Experimental): This is the intervention group that receives standard of care plus the WounDx™ report to augment the clinicians' judgment regarding the wounds readiness to close.
  Interventions: Device: Clinical Decision Support Tool

INTERVENTIONS:
Device: Clinical Decision Support Tool — WounDx is a clinical decision support tool that will help augment the clinicians' judgment regarding the wounds readiness to close.
  Other Names: WounDx
  Arms: WounDx
Procedure: Standard of Care (SOC) — The standard of care consists of serial wound irrigation, negative pressure wound therapy, and surgical debridement
  Other Names: Serial Wound Irrigation; Negative Wound Pressure Therapy; Surgical Debridement
  Arms: Standard of Care

SUMMARY:
The purpose of this research is to evaluate the overall use of the WounDx medical device in a clinical setting, such as a hospital. The WounDx device is experimental and not yet approved by the United States Food and Drug Administration (FDA). WounDx uses information about a patient's wound to generate a report that a surgeon may use to help determine when to close or not close the wound. The final decision to close the wound remains with the surgeon. The results from this pilot trial will inform a larger pivotal trial.

DETAILED DESCRIPTION:
Determining if a large, traumatic extremity wound is ready for successful delayed closure remains a challenge, as approximately 23%-25% of these wounds fail to heal after delayed closure is attempted, even when treated with aggressive surgical interventions, including debridement every 2-3 days. This pilot trial uses WounDx™, a device that aids clinicians in identifying extremity wounds that are likely to heal after surgical closure. The device is a Clinical Decision Support Tool (CDST) and consists of two main components: an immunoassay to obtain the expression of inflammatory biomarkers and, together with clinical data input, an interpretative algorithm. The purpose of the device is to identify wounds likely to proceed through normal phases of wound healing and, as a result, provide the clinician with a wound-specific prediction that an open traumatic extremity wound will heal successfully and remain closed if delayed closure is performed. The pilot trial serves as a proof of concept (POC) trial and establishes the overall feasibility of clinical operations (including recruitment, randomization, implementation of the intervention, and data collection). Trial enrollment is planned only for adults (≥18 to ≤65 years) with at least one traumatic extremity wound ≥75cm 2 , being treated with Negative Wound Pressure Therapy (NPWT), and delayed primary closure including split thickness skin grafting and rotational or free flaps. Local and systemic inflammatory biomarker expression will be assessed in wound effluent samples collected during subject treatment. These results will be input with other associated clinical data to WounDx™ to allow the device to provide a report including a recommendation on whether a specific wound should be closed within 48-72h of the previous debridement surgery, which is consistent with the current clinical practice guidelines. This pilot trial will inform the conduct of a larger, pivotal clinical trial to evaluate the safety and efficacy of WounDx™ in aiding clinicians identify traumatic extremity wounds ready for surgical closure.

ELIGIBILITY:
Inclusion Criteria:

* Wound surface area ≥75cm 2
* Extremity injury (including shoulder and buttock - without visceral communication)
* Wound amenable to Negative Pressure Wound Therapy using 3M™ V.A.C. ® canisters without gel pack

Exclusion Criteria:

* Insulin Dependent Diabetes
* Peripheral Vascular Disease
* Connective Tissue Disorders
* Preexisting immunosuppressive conditions or immunosuppression therapy
* Pregnancy
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of Patients from Each Site that Completes the Exploratory Outcome Measures | 1 year
  The primary outcome will be a report detailing the total number of patients from each site who have successfully completed all exploratory outcome measures. It is expected that a minimum of 3 patients from each site will complete required exploratory outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elster, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (5):
- United States (5):
  - University of Alabama - Birmingham Hospital, Birmingham, Alabama
  - Emory University / Grady Memorial Hospital, Atlanta, Georgia
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Duke University Hospital, Durham, North Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peoples GE, Jezior JR, Shriver CD. Caring for the wounded in Iraq--a photo essay. N Engl J Med. 2004 Dec 9;351(24):2476-80. doi: 10.1056/NEJMp048327. No abstract available. PMID 15622566
- [Background] Owens BD, Kragh JF Jr, Wenke JC, Macaitis J, Wade CE, Holcomb JB. Combat wounds in operation Iraqi Freedom and operation Enduring Freedom. J Trauma. 2008 Feb;64(2):295-9. doi: 10.1097/TA.0b013e318163b875. PMID 18301189
- [Background] Montgomery SP, Swiecki CW, Shriver CD. The evaluation of casualties from Operation Iraqi Freedom on return to the continental United States from March to June 2003. J Am Coll Surg. 2005 Jul;201(1):7-12; discussion 12-3. doi: 10.1016/j.jamcollsurg.2005.03.038. PMID 15978435
- [Background] Lisboa FA, Dente CJ, Schobel SA, Khatri V, Potter BK, Kirk AD, Elster EA. Utilizing Precision Medicine to Estimate Timing for Surgical Closure of Traumatic Extremity Wounds. Ann Surg. 2019 Sep;270(3):535-543. doi: 10.1097/SLA.0000000000003470. PMID 31348045